CLINICAL TRIAL: NCT04194151
Title: Impact of Propofol Dose Reduction in Relation to the Time Since Administration of Fentanyl During Anesthesia Induction
Brief Title: Impact of Propofol Reduction in Anesthesia Induction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Central de la Defensa Gómez Ulla (Other)
Responsible Party: Principal Investigator, paula agostina vullo, Sponsor-Investigator, Hospital Central de la Defensa Gómez Ulla
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 09/17
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Results first posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Propofol Adverse Reaction; Anesthesia
Keywords: propofol synergy; fentanyl; anesthesia induction
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Intervention Model Description: 2 time groups, divided into 3 dose groups
Who Masked: Participant
Masking Description: aleatory assignation, time measured by nurses, drugs administrated by principal investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 2 minute - 2 mg/kg group (Active Comparator): 2 mcg/kg of fentanyl administrated intravenously. wait for 2 minutes to inject 2 mg/kg of propofol
  Interventions: Drug: Propofol Injection
- 2 minute - 1,5 mg/kg group (Active Comparator): 2 mcg/kg of fentanyl administrated intravenously. wait for 2 minutes to inject 1,5 mg/kg of propofol
  Interventions: Drug: Propofol Injection
- 2 minute - 1 mg/kg group (Active Comparator): 2 mcg/kg of fentanyl administrated intravenously. wait for 2 minutes to inject 1 mg/kg of propofol
  Interventions: Drug: Propofol Injection
- 1 minute - 2 mg/kg group (Active Comparator): 2 mcg/kg of fentanyl administrated intravenously. wait for 1 minute to inject 2 mg/kg of propofol
  Interventions: Drug: Propofol Injection
- 1 minute - 1,5 mg/kg group (Active Comparator): 2 mcg/kg of fentanyl administrated intravenously. wait for 1 minute to inject 1,5 mg/kg of propofol
  Interventions: Drug: Propofol Injection
- 1 minute - 1 mg/kg group (Active Comparator): 2 mcg/kg of fentanyl administrated intravenously. wait for 1 minute to inject 1 mg/kg of propofol
  Interventions: Drug: Propofol Injection

INTERVENTIONS:
Drug: Propofol Injection — 1, 1.5 or 2 mg/kg of propofol according to the subgroup

SUMMARY:
Objective: Determine if, by reducing the dose of propofol and increasing the time elapsed between fentanyl and propofol administration, hemodynamic response is improved.

Methods: Patients were randomized into time groups (2 and 1 minute) and each subdivided into dose groups (1, 1.5 and 2 mg kg-1) obtaining six time-dose groups. After receiving 2 μg kg-1 of fentanyl, propofol was administered after the predetermined time. Time to hypnosis (BIS<60) and hemodynamic parameters at pre-induction, pre-intubation and postintubation were registered.

DETAILED DESCRIPTION:
A minimum of 162 patients were required, considering an expected Mean Difference of 5 with expected Standard Deviation of 22, confidence level of 95% and power of 80%. Estimating a possible loss of 15%, it was raised to 192. Consecutive identification numbers were assigned and the sample was randomized in six groups of 32 patients according to time and dose of propofol.

Pre-oxygenation was performed until the expired oxygen fraction exceeded 80% and 2 µg/kg of intravenous fentanyl were administered. Depending on the study group, 1 or 2 minutes were allowed to pass and 1, 1.5 or 2 mg/kg of propofol were supplied (prior administration of intravenous lidocaine 0.5 mg/kg). The time in which the BIS dropped below 60 was recorded. If it did not reach that level after two minutes or when it exceeded it but then rose above 60 again, an extra dose of propofol of 0.5 mg/kg was administered. Muscle relaxation was performed with rocuronium 0.6 mg/kg. The patient was manually ventilated until endotracheal intubation was performed by the same experienced anaesthesiologist and connected to mechanical ventilation.

Data were collected manually. Statistical analysis was performed using SPSS ver. 22. Inferential statistics were performed using t-test for quantitative variables, chi-square for qualitative and ANOVA for qualitative and quantitative comparisons. Non-parametric statistical tests were used when necessary. Confidence intervals were estimated at a level of 95% and a P value of <.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Adults who required general anesthesia
* General anesthesia with endotracheal intubation (no supraglottic devices)
* Signed informed consent
* Non-cardiac surgery
* Same anesthesiologist

Exclusion Criteria:

* Hemodynamic instability (systolic BP < 90 mmHg with clinical signs of low cardiac output: impaired consciousness, diuresis <0.5 ml/kg/h, central venous saturation <60% with normal arterial saturation or lactate >3 mmol/l)
* Increased risk of bronchoaspiration (absence of fasting, stomach retention, intestinal obstruction, pregnancy, etc.)
* Suspected difficult airway
* Known allergy to anesthetic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2018-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula A Vullo, MD, Principal Investigator
Locations (1):
- Hospital central de la defensa Gomez Ulla, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Every patient who agreed to participate and required general anesthesia with endotracheal intubation by the same anesthesiologist
Pre-assignment Details: Randomization was prior to data collection. The patient number was assigned by computerized randomizer to the 6 study groups. The collection was systematic from day one of the study, including all patients who met inclusion criteria and accepted participation.
  Of 192 patients enrolled, 186 met inclusion criteria.
Groups:
- 2 Minutes - 1 mg/kg Group: 2 mcg/kg of fentanyl administrated intravenously. wait for 2 minutes to inject 1 mg/kg of propofol
Period: Overall Study
Arm/Group | 2 Minute - 2 mg/kg Group | 2 Minute - 1,5 mg/kg Group | 2 Minutes - 1 mg/kg Group | 1 Minute - 2 mg/kg Group | 1 Minute - 1,5 mg/kg Group | 1 Minute - 1 mg/kg Group
Started | 32 | 32 | 32 | 32 | 32 | 32
Completed | 31 | 30 | 31 | 31 | 32 | 31
Not Completed | 1 | 2 | 1 | 1 | 0 | 1
Not completed — Physician Decision | 1 | 1 | 1 | 1 | 0 | 1
Not completed — Monitorization problem | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2 Minute - 2 mg/kg Group | 2 Minute - 1,5 mg/kg Group | 2 Minute - 1 mg/kg Group | 1 Minute - 2 mg/kg Group | 1 Minute - 1,5 mg/kg Group | 1 Minute - 1 mg/kg Group | Total
Number analyzed (Participants) | 31 | 30 | 31 | 31 | 32 | 31 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (20) | 61 (17) | 60 (19) | 59 (17) | 64 (18) | 55 (16) | 60 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 17 | 17 | 18 | 14 | 95
  Male | 16 | 16 | 14 | 14 | 14 | 17 | 91
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
weight [Mean (Standard Deviation); unit: kilograms] | 73 (16) | 77 (17) | 70 (15) | 71 (15) | 71 (15) | 73 (15) | 72 (15)
anesthesia risk (ASA), categorical [Count of Participants; unit: Participants] — Low risk: ASA I-II High risk: ASA III-IV
  Participants
    Low risk | 20 | 19 | 17 | 21 | 13 | 21 | 111
    High risk | 11 | 11 | 14 | 10 | 19 | 10 | 75
Hypertension [Count of Participants; unit: Participants] | 15 | 9 | 15 | 13 | 16 | 13 | 81
Antihypertensive treatment [Count of Participants; unit: Participants] | 9 | 9 | 12 | 10 | 12 | 11 | 63
Heart rate treatment [Count of Participants; unit: Participants] — B-Blockers or Calcium antagonists
  Participants | 11 | 7 | 10 | 9 | 11 | 3 | 51

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure Variation
Description: Non-invasive systolic blood pressure change (%) at baseline, pre-intubation and postintubation. Positive results mean percentage reduction in SBP between the studied moments. Negative results mean percentage increase in SBP between the studied moments.
Time Frame: Baseline before fentanyl administration, pre-intubation after propofol and bispectral index<60 and postintubation 15 seconds after endotracheal tube positioned
Measure: Mean (Standard Deviation); unit: percentage of variation
Arm/Group | 2 Minute - 2 mg/kg Group | 2 Minute - 1,5 mg/kg Group | 2 Minute - 1 mg/kg Group | 1 Minute - 2 mg/kg Group | 1 Minute - 1,5 mg/kg Group | 1 Minute - 1 mg/kg Group
Number analyzed (Participants) | 31 | 30 | 31 | 31 | 32 | 31
percentage of variation
  SBP baseline/pre-intubation | 26 (16) | 23 (12) | 18 (13) | 22 (11) | 18 (13) | 17 (13)
  SBP baseline/postintubation | 11 (22) | 8 (15) | 9 (19) | 14 (18) | 16 (19) | 8 (16)
  SBP pre-intubation/postintubation | -22 (27) | -21 (28) | -12 (17) | -12 (21) | -3 (16) | -12 (16)

2. Primary Outcome: Heart Rate Variation
Description: Heart rate change (%) registered at baseline, pre-intubation and postintubation. Positive results mean percentage reduction in HR between the studied moments. Negative results mean percentage increase in HR between the studied moments.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of variation
Arm/Group | 2 Minute - 2 mg/kg Group | 2 Minute - 1,5 mg/kg Group | 2 Minute - 1 mg/kg Group | 1 Minute - 2 mg/kg Group | 1 Minute - 1,5 mg/kg Group | 1 Minute - 1 mg/kg Group
Number analyzed (Participants) | 31 | 30 | 31 | 31 | 32 | 31
percentage of variation
  HR baseline/pre-intubation | 6 (13) | 4 (8) | 4 (10) | 1 (11) | 4 (15) | 5 (14)
  HR baseline/postintubation | -10 (19) | -8 (15) | -9 (16) | -4 (17) | -5 (20) | -10 (18)
  HR pre-intubation/postintubation | -17 (19) | -12 (16) | -15 (20) | -5 (16) | -10 (19) | -17 (19)

3. Primary Outcome: Systolic Blood Pressure Variation in Elderly (>55y)
Description: Non-invasive SBP change (%) in patients > 55 years at baseline, pre-intubation and postintubation. Positive results mean percentage reduction in SBP between the studied moments. Negative results mean percentage increase in SBP between the studied moments.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of variation
Arm/Group | 2 Minute - 2 mg/kg Group | 2 Minute - 1,5 mg/kg Group | 2 Minute - 1 mg/kg Group | 1 Minute - 2 mg/kg Group | 1 Minute - 1,5 mg/kg Group | 1 Minute - 1 mg/kg Group
Number analyzed (Participants) | 18 | 23 | 18 | 16 | 21 | 13
percentage of variation
  SBP baseline/pre-intubation | 36 (12) | 26 (12) | 21 (13) | 29 (6) | 21 (13) | 22 (13)
  SBP baseline/postintubation | 19 (22) | 10 (14) | 13 (19) | 22 (15) | 22 (17) | 12 (13)
  SBP pre-intubation/postintubation | -27 (32) | -23 (30) | -10 (16) | -10 (23) | 2 (13) | -15 (19)

4. Secondary Outcome: Time to Hypnosis
Description: Bispectral index (BIS)<60 meaning "general anesthesia", BIS>60 meaning mild/moderate sedation. We measure the time until patient reachs hypnosis
Time Frame: After administration of propofol, time is measured in seconds until BIS values are less than 60
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | 2 Minute - 2 mg/kg Group | 2 Minute - 1,5 mg/kg Group | 2 Minute - 1 mg/kg Group | 1 Minute - 2 mg/kg Group | 1 Minute - 1,5 mg/kg Group | 1 Minute - 1 mg/kg Group
Number analyzed (Participants) | 31 | 30 | 31 | 31 | 32 | 31
seconds | 54 (29) | 49 (27) | 62 (34) | 41 (20) | 47 (15) | 67 (42)

5. Secondary Outcome: Number of Patients Who Needed Vasoactive Drug
Description: Patients who suffered SPB reduction > 30% or SPB < 90mmHg, receive vasoactive drugs
Time Frame: 1 minute after intubation
Measure: Count of Participants; unit: Participants
Arm/Group | 2 Minute - 2 mg/kg Group | 2 Minute - 1,5 mg/kg Group | 2 Minute - 1 mg/kg Group | 1 Minute - 2 mg/kg Group | 1 Minute - 1,5 mg/kg Group | 1 Minute - 1 mg/kg Group
Number analyzed (Participants) | 31 | 30 | 31 | 31 | 32 | 31
Participants | 4 | 1 | 0 | 2 | 3 | 0

ADVERSE EVENTS:
Time Frame: Baseline until 60 seconds after endotracheal tube positioned
Description: Extreme bradicardia (HR<40) Extreme hypotension (SBP <60)
Arm/Group | 2 Minute - 2 mg/kg Group | 2 Minute - 1,5 mg/kg Group | 2 Minute - 1 mg/kg Group | 1 Minute - 2 mg/kg Group | 1 Minute - 1,5 mg/kg Group | 1 Minute - 1 mg/kg Group
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30 | 0/31 | 0/31 | 0/32 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30 | 0/31 | 0/31 | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 4/31 | 1/30 | 0/31 | 2/31 | 3/32 | 0/31
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 Minute - 2 mg/kg Group (N=31) | 2 Minute - 1,5 mg/kg Group (N=30) | 2 Minute - 1 mg/kg Group (N=31) | 1 Minute - 2 mg/kg Group (N=31) | 1 Minute - 1,5 mg/kg Group (N=32) | 1 Minute - 1 mg/kg Group (N=31)
Vasoactive drug need (Cardiac disorders) | 4 (4) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0) — SBP reduction >30% or SBP < 90mmHg

LIMITATIONS AND CAVEATS:
Pediatric population not included. BMI not registrated. Type of surgery not registered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/51/NCT04194151/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/51/NCT04194151/Prot_SAP_001.pdf